CLINICAL TRIAL: NCT02815189
Title: Incidence of Flare-ups and Apical Healing After Single-visit or Two-visits Treatment of Teeth With Necrotic Pulp and Apical Periodontitis After a Two-year Control Period. A Randomised Clinical Trial.
Brief Title: Incidence of Flare-ups and Apical Healing After Single-visit or Two-visits Treatment.
Acronym: FlareUp
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universidad Autonoma de Baja California (Other)
Responsible Party: Principal Investigator, Jorge Paredes Vieyra, DDS, MsC, PhD, Universidad Autonoma de Baja California
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 52016
Record Dates: First submitted 2016-06-02; First posted 2016-06-28 (Estimated); Last update posted 2017-05-02 (Actual); Status verified 2017-05

CONDITIONS: Pain
Keywords: pain
MeSH Terms: conditions — Pain | interventions — Ibuprofen; Dental Implantation, Endosseous, Endodontic; Acetaminophen

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Post operative Pain after a RCT (Experimental): Ibuprofen for Post operative pain. Take 400 mg taken a week after. Incidence of flare ups after a single vs multiple visits root canal treatments.
  Interventions: Procedure: Ibuprofen for post operative pain; Drug: Acetaminophen 325 mg for Flare up
- Flare up (Experimental): Acetaminophen 325 mg for Flare Up. Taken second day after. Incidence of Post operative pain after root canal treatment in one vs two visits.
  Interventions: Procedure: Ibuprofen for post operative pain; Drug: Acetaminophen 325 mg for Flare up

INTERVENTIONS:
Procedure: Ibuprofen for post operative pain — All treatment sessions were approximately 50 minutes in length to allow for acceptable time for completion of treatment and retreatment in one or two visits. All the clinical procedures were performed by the author. Following local anesthesia with 2% lidocaine with 1:100,000 epinephrine (Septodont Saint-Maur des Fossés, France) and rubber dam isolation the tooth was disinfected with 5.25% NaOCl (Ultra bleach, Bentonville, AR, USA).
  Other Names: Endodontic therapy
Drug: Acetaminophen 325 mg for Flare up — Each patient will be evaluated a week after completion the clinical procedures.
  Other Names: Endodontic procedures

SUMMARY:
Aim to compare Incidence of flare-ups and apical healing after single-visit or two-visits treatment of teeth with necrotic pulp and apical periodontitis after a two-year control period.

110 teeth with a diagnosis of pulp necrosis and apical radiolucency at the apex. Working length was established with EAL and confirmed radiographically. M4 system with Flex-R files were used to complete canal preparation. Level of discomfort were recorded and cases with severe postoperative pain and/or swelling were classified as flare-ups.

DETAILED DESCRIPTION:
110 teeth with a diagnosis of pulp necrosis and apical radiolucency at the apex. Working length was established with EAL and confirmed radiographically. M4 system with Flex-R files were used to complete canal preparation. Level of discomfort were recorded and cases with severe postoperative pain and/or swelling were classified as flare-ups.

ELIGIBILITY:
Inclusion Criteria:

* a) Radiographic evidence of apical periodontitis (minimum size ≥2.0 mm x 2.0 mm) and a diagnosis of pulpal necrosis confirmed by negative response to hot and cold tests and b) Need for retreatment. Thermal pulp testing was performed by the author, and radiographic interpretation was verified by one certified oral surgeon.

Exclusion Criteria:

* patients without inclusion requirements or failure to obtain patient´s authorization. Patients, were excluded if they were younger than 18 years old, pregnant, had a positive history of antibiotic use within the past month, suffered from diabetes, or other systemic diseases. Teeth with periodontal pockets deeper than 4 mm also were excluded of the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2014-02; Primary Completion 2016-02 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
Pain intensity measure with general pain scale | a week
  Each patient will recall a week to evaluate post operative pain

CONTACTS AND LOCATIONS:
Overall Officials: Miguel O Millan, PhD, Study Chair — Mexico: Secretaria de Salud

IPD SHARING:
Plan to Share IPD: Yes
Each participant will be evaluated a week after the treatment.